CLINICAL TRIAL: NCT07080034
Title: A Randomized Double-Blind, Placebo-Controlled Study of the Efficacy, Safety, Pharmacokinetics, Pharmacodynamics, and Immunogenicity of BCD-261 in Subjects With Moderate to Severe Active Ulcerative Colitis
Brief Title: Study of the Efficacy, Safety, Pharmacokinetics, Pharmacodynamics, and Immunogenicity of BCD-261 in Subjects With Moderate to Severe Active Ulcerative Colitis
Acronym: ULTRAMARINE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Biocad (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BCD-261-4
Record Dates: First submitted 2025-07-15; First posted 2025-07-23 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Ulcerative Colitis (UC)
Keywords: biologics; ulcerative colitis; monoclonal antibodies; TL1A
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- BCD-261, medium dose induction/ low dose maintenance regimens (Experimental): Group 1: Subjects in this arm will receive a medium dose of the BCD-261 subcutaneously once every 4 weeks until Week 12 during the induction regimen (Weeks 0-12), followed by a transition to a maintenance regimen with a low dose of the BCD-261 once every 8 weeks from Week 20 to Week 100.
  Interventions: Biological: anti-TL1A monoclonal antibody, low dose; Biological: anti-TL1A monoclonal antibody, medium dose
- BCD-261, medium dose induction/ medium dose maintenance regimens (Experimental): Group 2: Subjects in this arm will receive a medium dose of the BCD261 subcutaneously once every 4 weeks until Week 12 during the induction regimen (Weeks 0-12), followed by the maintenance regimen with the same dose of the BCD-261 once every 8 weeks from Week 20 to Week 100.
  Interventions: Biological: anti-TL1A monoclonal antibody, medium dose
- BCD-261, high dose induction/ medium dose maintenance regimens (Experimental): Group 3: Subjects in this arm will receive a high dose of the BCD-261 subcutaneously once every 4 weeks until Week 12 during the induction regimen (Weeks 0-12) , followed by a transition to a maintenance regimen with a medium dose of the BCD-261 once every 8 weeks from Week 20 to Week 100.
  Interventions: Biological: anti-TL1A monoclonal antibody, medium dose; Biological: anti-TL1A monoclonal antibody, high dose
- BCD-261, high dose induction/ high dose maintenance regimens (Experimental): Group 4: Subjects in this arm will receive a high dose of the BCD261 subcutaneously once every 4 weeks until Week 12 during the induction regimen (Weeks 0-12), followed by maintenance regimen with with the same dose of the BCD-261 once every 8 weeks from Week 20 to Week 100.
  Interventions: Biological: anti-TL1A monoclonal antibody, high dose
- Placebo (Placebo Comparator): Group 5: Subjects in this arm will receive placebo subcutaneously at Weeks 0, 4, 8, and 12, followed by a medium dose of the BCD-261 subcutaneously once every 4 weeks until Week 28 , followed by a transition to a low dose of the BCD-261 once every 8 weeks from Week 36 to Week 100.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: anti-TL1A monoclonal antibody, low dose — injection
  Arms: BCD-261, medium dose induction/ low dose maintenance regimens
Biological: anti-TL1A monoclonal antibody, medium dose — injection
  Arms: BCD-261, high dose induction/ medium dose maintenance regimens; BCD-261, medium dose induction/ low dose maintenance regimens; BCD-261, medium dose induction/ medium dose maintenance regimens
Biological: anti-TL1A monoclonal antibody, high dose — injection
  Arms: BCD-261, high dose induction/ high dose maintenance regimens; BCD-261, high dose induction/ medium dose maintenance regimens
Other: Placebo — injection
  Arms: Placebo

SUMMARY:
The aim of the study is to evaluate the efficacy, safety, pharmacokinetics, pharmacodynamics and immunogenicity of study drug (BCD-261) in comparison with placebo and to characterize the dose-response relationship in patients with moderate to severe active ulcerative colitis. The study will be conducted in a population of male and female subjects ≥18 years and ≤75 years with moderate to severe active ulcerative colitis and an inadequate response to prior treatment with glucocorticoids, immunosuppressants, or biologics/targeted immunosuppressants.

DETAILED DESCRIPTION:
Subjects meeting the eligibility criteria will be randomized in 5 groups to receive one of four studied dosage regimens of BCD-261 or placebo. The study groups will differ in drug dosages of BCD-261 (low, medium, high) during the induction and maintenance periods of therapy. After the primary endpoint assessment subjects in placebo group will be switched to BCD-261 medium studied dose.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of ulcerative colitis with involvement of the colon proximal to the rectum (≥15 cm from the distal edge of the anal canal), established ≥3 months before signing the ICF and confirmed by endoscopic examination data.

2. Moderate to severe active ulcerative colitis with a modified Mayo score (mMS) of ≥4 and ≤9 points, which includes an endoscopic component of ≥2 points (according to a central independent review) and a stool blood score of ≥1 point.

3. Inadequate response to therapy according to the investigator's assessment, manifested by at least one of the following signs:

1. Persistent symptoms of disease activity despite treatment with at least one course of glucocorticoids including prednisolone at a dose of ≥40 mg/day or equivalent or budesonide ≥9 mg/day or equivalent for at least 2 weeks with oral administration (at least 1 week with intravenous administration at a dose equivalent to oral prednisolone ≥40 mg/day).
2. Steroid dependence manifested by an increase in disease activity after initial improvement, with a decrease in the dose of glucocorticoids below the dose equivalent to 10 mg of oral prednisolone per day, within 3 months from the beginning of treatment, or a relapse of the disease within 3 months after the end of glucocorticoid use.
3. Persistent symptoms of disease activity despite treatment with at least one course of immunosuppressants (azathioprine at a dose of ≥2.0 mg/kg and/or 6-mercaptopurine at a dose of ≥1.0 mg/kg) for ≥12 weeks, or in response to another treatment regimen with these drugs according to a regional standard of care.
4. Primary lack of response to therapy with TNFa inhibitors and/or anti-integrins, and/or IL-12/23 inhibitors, and/or Janus kinase inhibitors, and/or sphingosine-1-phosphate receptor modulators, defined as the persistence of symptoms of disease activity despite at least one course of induction of remission according to a treatment scheme approved by the regional standard.
5. Loss of response to therapy with TNFa inhibitors and/or anti-integrins, and/or IL-12/23 inhibitors, and/or Janus kinase inhibitors, and/or sphingosine-1-phosphate receptor modulators, defined as the appearance of symptoms of disease activity after initial improvement as a result of treatment with at least one course of induction of remission and at least one course of maintenance of remission according to a treatment scheme approved by the regional standard.
6. A history of intolerance to glucocorticoids and/or immunosuppressants (azathioprine, 6-mercaptopurine) and/or biological therapy/targeted immunosuppressants (TNFa inhibitors, anti-integrins, anti-IL-12/23 monoclonal antibodies, Janus kinase inhibitors, sphingosine-1-phosphate receptor modulators) established by the treating physician.

4. Maintaining a stable dose of concomitant medications for ≥2 weeks prior to signing the ICF and in the screening period for glucocorticoids and 5-ASCs and for ≥4 weeks prior to signing the ICF and in the screening period for immunosuppressants (azathioprine, 6-mercaptopurine).

Exclusion Criteria:

1. A history of or current at the time of signing the ICF Crohn's disease, unspecified colitis, ischemic colitis, radiation colitis, microscopic colitis, complicated form of diverticular disease.
2. A history of primary sclerosing cholangitis.
3. A history of fulminant colitis, toxic dilation of the colon, intestinal obstruction, intestinal perforation (except for those caused by injury or appendicitis).
4. A history of dysplasia of any grade in any part of the gastrointestinal tract at the time of signing the ICF.
5. Presence of intestinal stoma or artificial rectum or the need for them.
6. Failure of ≥3 classes of biologics/targeted immunosuppressors (according to INN) with different mechanisms of action (TNFa inhibitors, anti-integrins, IL-12/23 inhibitors, Janus kinase inhibitors, sphingosine-1-phosphate receptor modulators) or ≥4 biologics/targeted immunosuppressants, regardless of the mechanism of action.
7. Use of any of the indicated therapies within the specified time frame or need for therapy with these drugs during the study period:

(1) Use of Janus kinase inhibitors within 2 weeks prior to signing the ICF or during the screening period.

(2) Use of TNFa inhibitors within 8 weeks prior to signing the ICF or during the screening period.

(3) Using modulators of sphingosine-1-phosphate receptors within 10 weeks prior to signing the ICF or during the screening period.

(4) Use of anti-integrins, IL-12/23 inhibitors within 12 weeks before signing the ICF or during the screening period.

(5) Use of oral glucocorticoids at a dose equivalent to prednisone >20 mg/day or budesonide >9 mg/day or rectal administration of glucocorticoids at any dose within

2 weeks prior to signing the ICF or during the screening period or parenteral administration of glucocorticoids at any dose within 4 weeks prior to signing the ICF or during the screening period.

(6) Rectal administration of 5-ASCs within 2 weeks prior to signing the ICF or during the screening period.

(7) Use of immunosuppressants not included in the approved therapy (tacrolimus, cyclosporine, mycophenolate mofetil, rapamycin, leflunomide, penicillamine, etc.) within 4 weeks before signing the ICF or during the screening period.

(8) Long-term regular use of non-steroidal anti-inflammatory drugs (≥3 times a week for ≥6 weeks) for 2 weeks prior to signing the ICF.

(9) Use of any other investigational drugs in other clinical trials at the time of signing the ICF or less than 8 weeks or 5 half-lives (whichever is longer) before the date of randomization.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Estimated)
Dates: Start 2025-08-14 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects who achieved clinical remission | week 14
  Proportion of subjects with modified Mayo score ≤2 points (endoscopic mucosal score ≤1, stool blood score = 0, stool frequency score ≤1, assessment for each component should not exceed the baseline level)

SECONDARY OUTCOMES:
Proportion of subjects who achieved clinical remission | week 24
  Proportion of subjects with modified Mayo score ≤2 points (endoscopic mucosal score ≤1, stool blood score = 0, stool frequency score ≤1, assessment for each component should not exceed the baseline level)

OTHER OUTCOMES:
Proportion of subjects who achieved a clinical response | weeks 14, 24, 52, 100
  Proportion of subjects modified Mayo score of ≥2 points and ≥30% from the baseline with a decrease in the estimated stool blood score of ≥1 point from the baseline or the estimated stool blood score of ≤1 point)
Proportion of subjects who achieved clinical remission | weeks 52, 100
  Proportion of subjects with modified Mayo score ≤2 points (endoscopic mucosal score ≤1, stool blood score = 0, stool frequency score ≤1, assessment for each component should not exceed the baseline level)
Proportion of subjects who achieved clinical remission | weeks 24, 52, 100
  Proportion of subjects with modified Mayo score ≤2 points (endoscopic mucosal score ≤1, stool blood score = 0, stool frequency score ≤1, assessment for each component should not exceed the baseline level) among subjects who had a clinical response according to the modified Mayo score at Week 14
Proportion of subjects who achieved clinical remission | weeks 52, 60, 100
  Proportion of subjects with modified Mayo score ≤2 points (endoscopic mucosal score ≤1, stool blood score = 0, stool frequency score ≤1, assessment for each component should not exceed the baseline level) without the use of glucocorticoids (for at least 12 weeks) among subjects who initially received glucocorticoid therapy
Proportion of subjects who achieved clinical remission | weeks 14, 24, 52, 100
  Proportion of subjects with Mayo score of ≤2 (each component of the score ≤1, but not higher than the baseline)
Proportion of subjects who achieved an endoscopic response | weeks 14, 24, 52, 100
  Proportion of subjects with mucosal state assessment according to the Mayo endoscopic score of ≤1 without friability. Mayo Endoscopic Score (MES) is a widely used tool for assesing the stage of ulcerative colitis based solely on endoscopic examination. MES may vary from 0 to 3, where 0 corresponds to normal or inactive, 1 - to mild, 2- to moderate and 3 - to severe disease activity.
Proportion of subjects who achieved endoscopic remission (mucosal healing) | weeks 14, 24, 52, 100
  Proportion of subjects with a Mayo endoscopic score of 0. Mayo Endoscopic Score (MES) is a widely used tool for assesing the stage of ulcerative colitis based solely on endoscopic examination. MES may vary from 0 to 3, where 0 corresponds to normal or inactive, 1 - to mild, 2- to moderate and 3 - to severe disease activity.
Proportion of subjects who achieved an endoscopic and histological response | weeks 14, 24, 52, 100
  Proportion of subjects with Mayo endoscopic score of ≤1 without friability in combination with a Geboes score ≤3.1. Mayo Endoscopic Score (MES) is a widely used tool for assesing the stage of ulcerative colitis based solely on endoscopic examination. MES may vary from 0 to 3, where 0 corresponds to normal or inactive, 1 - to mild, 2- to moderate and 3 - to severe disease activity. Histologic Geboes Score is the most commonly used histological score in ulcerative colitis. Evaluation according to the histologic Geboes score is divided into 6 grades: architectural changes [grade 0], chronic inflammatory infiltrate [grade 1], lamina propria neutrophils and eosinophils [grade 2], neutrophils in epithelium [grade 3], crypt destruction [grade 4] and erosions or ulcerations [grade 5], and each grade of the score is divided in 4 subcategories. The Geboes score ranges from 0.0 to 5.4, with higher values indicating more severe inflammation.
Change in the Geboes score from the baseline. | weeks 14, 24, 52, 100
  Evaluation according to the histologic Geboes score is divided into 6 grades: architectural changes [grade 0], chronic inflammatory infiltrate [grade 1], lamina propria neutrophils and eosinophils [grade 2], neutrophils in epithelium [grade 3], crypt destruction [grade 4] and erosions or ulcerations [grade 5], and each grade of the score is divided in 4 subcategories. The Geboes score ranges from 0.0 to 5.4, with higher values indicating more severe inflammation.
Change in the partial Mayo score from the baseline | weeks 14, 24, 52, 100
  The assessment of the partial Mayo score ranges from 0 to 9 points, which are derived from 3 subscores, each of which is evaluated as 0 to 3 points:
  * Stool frequency assessment (0 to 3 points).
  * Evaluation of blood presence in the stool (0 to 3 points).
  * Physician's global assessment (0 to 3 points). A higher score indicates greater disease activity. It is a modification of the total Mayo score, from which Mayo Endoscopic Score (MES) was excluded.
Proportion of subjects who achieved a clinical response of ≥50% from baseline | weeks 14, 24, 52, 100
  Clinical response measured by two-component patient reported outcomes (PRO2) scale consist of the patient-derived items from the Mayo score (rectal bleeding and stool frequency). PRO2 scale ranges from 0-6 with higher values indicating worse outcome.
Change in the fecal calprotectin level from the baseline | weeks 14, 24, 52, 100
Change in the highly sensitive C-reactive protein level from the baseline | weeks 14, 24, 52, 100
Changes in the proportion of subjects with extra-intestinal manifestations from the baseline | weeks 14, 24, 52, 100.

CONTACTS AND LOCATIONS:
Overall Officials: Arina V Zinkina-Orikhan, Study Director — Director of Clinical Development Department, BIOCAD
Locations (19):
- Russia (19):
  - LLC Medical Center "ASTRA", Barnaul, Altayskiy Kray
  - Republican Clinical Hospital named after G.G. Kuvatov, Ufa, Bashkortostan Republic
  - Federal State Educational Institution of Higher Education "Rostov State Medical University" of the Ministry of Health of the Russian Federation, Rostov-on-Don, Rostov Oblast
  - State Autonomous Institution of Healthcare "Republican Clinical Hospital of the Ministry of Healthcare of the Republic of Tatarstan", Kazan', Tatarstan Republic
  - "South Ural State Medical University" of the Ministry of Health of the Russian Federation, Chelyabinsk
  - Federal Siberian Scientific and Clinical Center of the Federal Medical and Biological Agency, Krasnoyarsk
  - Regional State Healthcare Institution "Regional Clinical Hospital", Krasnoyarsk
  - Llc "Olla-Med", Moscow
  - Moscow Clinical Scientific and Practical Center named after A.S. Loginov of the Moscow City Health Department, Moscow
  - State Healthcare Institution of the City of Moscow "V.M. Buyanov City Clinical Hospital of the Moscow City Healthcare Department", Moscow
  - Branch of the LLC "Hadassah Medical LTD", Moscow
  - State Institution of Healthcare of the Moscow Region "Moscow Regional Research Clinical Institute named after M.F. Vladimirsky", Moscow
  - Llc "Novosibirsk Gastrocenter", Novosibirsk
  - Federal State Educational Institution of Higher Education "North-West State Medical University named after I.I. Mechnikov" of the Ministry of Health of the Russian Federation, Saint Petersburg
  - Saint Petersburg State Healthcare Institution "City Hospital of the Holy Martyr Elizabeth", Saint Petersburg
  - Federal State Educational Institution of Higher Education "First Saint Petersburg State Medical University named after Academician I.P. Pavlov" of the Ministry of Health of the Russian Federation, Saint Petersburg
  - LLC "Research Center Eco-Safety", Saint Petersburg
  - State Healthcare Institution Ulyanovsk Regional Clinical Hospital, Ulyanovsk
  - State Healthcare Institution "Primorsky Regional Clinical Hospital No. 1", Vladivostok

IPD SHARING:
Plan to Share IPD: No